CLINICAL TRIAL: NCT00095511
Title: A Multicenter, Randomized, Double-Blind, Placebo Controlled Study of Aripiprazole Monotherapy in the Treatment of Acutely Manic Patients With Bipolar I Disorder
Brief Title: Aripiprazole in Patients With Acute Mania
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka America Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CN138-135
Record Dates: First submitted 2004-11-05; First posted 2004-11-08 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2008-05

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Mania
MeSH Terms: conditions — Bipolar Disorder | interventions — Aripiprazole

INTERVENTIONS:
Drug: aripiprazole

SUMMARY:
The purpose of this trial is to test the safety & efficacy of aripiprazole in patients with Bipolar Mania for a period of at least 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Acute Bipolar I Mania

Exclusion Criteria:

* Patients with a DSM-IV diagnosis other than Bipolar I Mania

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 615
Dates: Start 2004-06; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline to endpoint in a mania rating scale

SECONDARY OUTCOMES:
Response rate and Clinical Global Impression scale at endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (38):
- United States (38):
  - Local Institution, Tuscaloosa, Alabama
  - Local Institution, Scottsdale, Arizona
  - Local Institution, Cerritos, California
  - Local Institution, Garden Grove, California
  - Local Institution, La Palma, California
  - Local Institution, Riverside, California
  - Local Institution, San Diego, California
  - Local Institution, Denver, Colorado
  - Local Institution, Middletown, Connecticut
  - Local Institution, New Haven, Connecticut
  - Local Institution, Bradenton, Florida
  - Local Institution, Kissimmee, Florida
  - Local Institution, Maitland, Florida
  - Local Institution, Augusta, Georgia
  - Local Institution, Honolulu, Hawaii
  - Local Institution, Chicago, Illinois
  - Local Institution, Hoffman Estates, Illinois
  - Local Institution, Indianapolis, Indiana
  - Local Institution, Louisville, Kentucky
  - Local Institution, New Orleans, Louisiana
  - Local Institition, Shreveport, Louisiana
  - Local Institution, Saint Charles, Missouri
  - Local Institution, Clementon, New Jersey
  - Local Institution, Cedarhurst, New York
  - Local Institution, Elmsford, New York
  - Local Institution, Holliswood, New York
  - Local Institution, Morganton, North Carolina
  - Local Institution, Raleigh, North Carolina
  - Local Institution, Cincinnati, Ohio
  - Local Institution, Cleveland, Ohio
  - Local Institution, Lyndhurst, Ohio
  - Local Institution, Oklahoma City, Oklahoma
  - Local Institution, Norristown, Pennsylvania
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Austin, Texas
  - Local Institution, Bellaire, Texas
  - Local Institution, Houston, Texas
  - Local Institution, Arlington, Virginia

REFERENCES:
- [Background] Keck PE, Orsulak PJ, Cutler AJ, Sanchez R, Torbeyns A, Marcus RN, McQuade RD, Carson WH; CN138-135 Study Group. Aripiprazole monotherapy in the treatment of acute bipolar I mania: a randomized, double-blind, placebo- and lithium-controlled study. J Affect Disord. 2009 Jan;112(1-3):36-49. doi: 10.1016/j.jad.2008.05.014. Epub 2008 Oct 2. PMID 18835043
- [Derived] McIntyre RS, McElroy SL, Eudicone JM, Forbes RA, Carlson BX, Baker RA. A 52-week, double-blind evaluation of the metabolic effects of aripiprazole and lithium in bipolar I disorder. Prim Care Companion CNS Disord. 2011;13(6):PCC.11m01182. doi: 10.4088/PCC.11m01182. PMID 22454801